CLINICAL TRIAL: NCT07195773
Title: Effects of Repetitive Transcranial Magnetic Stimulation on Corticomotor Excitability and Balance Performance in People With Parkinson's Disease
Brief Title: Effects of rTMS on Corticomotor Excitability and Balance Performance in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CS2-23200
Record Dates: First submitted 2024-05-07; First posted 2025-09-29 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Parkinson Disease; Motor Cortex; Excitability; Balance; Motor Skills Disorders
MeSH Terms: conditions — Parkinson Disease; Motor Skills Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): Patients in this group first undergo high-frequency rTMS treatment, followed by a two-week rest period, then proceed to low-frequency rTMS after another two-week rest, and finally receive sham stimulation rTMS.
  rTMS high-frequency 1Hz 80%RMT rTMS low-frequency 1Hz 80%RMT rTMS sham 10HZ 20%RMT
  Interventions: Device: rTMS
- Group B (Experimental): Patients in this group first undergo low-frequency rTMS treatment, followed by a two-week rest period, then proceed to high-frequency rTMS after another two-week rest, and finally receive sham stimulation rTMS.
  rTMS high-frequency 1Hz 80%RMT rTMS low-frequency 1Hz 80%RMT rTMS sham 10HZ 20%RMT
  Interventions: Device: rTMS
- Group C (Experimental): Patients in this group first undergo sham stimulation rTMS treatment, followed by a two-week rest period, then proceed to high-frequency rTMS after another two-week rest, and finally receive low-frequency rTMS.
  rTMS high-frequency 1Hz 80%RMT rTMS low-frequency 1Hz 80%RMT rTMS sham 10HZ 20%RMT
  Interventions: Device: rTMS

INTERVENTIONS:
Device: rTMS — investigate the effects of repetitive transcranial magnetic stimulation on corticomotor excitability, balance performance, and mobility in patients with Parkinson's disease, and to further explore the effects on corticomotor excitability by single low-frequency and high-frequency repetitive transcranial magnetic stimulation. Participants will receive different stimulation approaches in sequences: high-frequency rTMS, low-frequency rTMS, and sham rTMS. They will be randomly assigned to three groups with different stimulation sequences. After each single stimulation, corticomotor excitability, balance, and motor symptoms will be measured. In this study, eighteen PD patients with Hoehn and Yahr stage 1 to 3 will be recruited.

SUMMARY:
The study investigates the effects of repetitive transcranial magnetic stimulation on motor cortex excitability, balance, and motor function in patients with Parkinson's disease. Additionally, it further examines the effects of single-session low-frequency and high-frequency repetitive transcranial magnetic stimulation on motor cortex excitability.

DETAILED DESCRIPTION:
The study investigates the effects of repetitive transcranial magnetic stimulation on motor cortex excitability, balance, and motor function in patients with Parkinson's disease. Additionally, it further examines the effects of single-session low-frequency and high-frequency repetitive transcranial magnetic stimulation on motor cortex excitability.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with primary Parkinson's disease
2. Age: 40-85 years
3. Hoehn and Yahr scale (H&Y scale) : I-III
4. Appropriate prescribed medication, and regular intake for more than 2 weeks
5. Can walk more than 10m with or without the use of assistive devices

Exclusion Criteria:

1. Any other neurological presentation (Excluding PD)
2. Any neurological surgery that would affect participation in this experiment
3. Orthopedic pathology and Cardiovascular issues
4. MMSE≦24
5. Exercise used for treatment in the last three months
6. Contraindications for transcranial magnetic stimulation (Presence of metal implants in the head and neck, a pacemaker in the chest, personal or family history of epilepsy, recent brain injury, currently taking antidepressant medication.)

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2024-12-16 (Actual); Primary Completion 2025-11-19 (Actual); Study Completion 2025-11-19 (Actual)

PRIMARY OUTCOMES:
Cortical excitability | Cortical excitability will be assessed before and immediately after each intervention. Each intervention is separated by a 2-week washout period. All assessments occur within an 4-week period.
  Transcranial magnetic stimulation
Motor function | UPDRS-III will be assessed before and immediately after each intervention. Each intervention is separated by a 2-week washout period. All assessments occur within an 4-week period.
  UPDRS-III

SECONDARY OUTCOMES:
Dynamic balance | FRT will be assessed before and immediately after each intervention. Each intervention is separated by a 2-week washout period. All assessments occur within an 4-week period.
  Functional Reach Test
Functional mobility | TUG will be assessed before and immediately after each intervention. Each intervention is separated by a 2-week washout period. All assessments occur within an 4-week period.
  Timed Up and Go test

CONTACTS AND LOCATIONS:
Overall Officials: LIU HSIN-HSUAN, PhD, Study Chair — Assistant Professor; HONG SONG-PING, BSc, Principal Investigator — student
Locations (1):
- Chung Shan Medical Unirversity, Taichung, Southern District, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
The purpose of the first study is to investigate the effects of repetitive transcranial magnetic stimulation on corticomotor excitability, balance performance, and mobility in patients with Parkinson's disease, and to further explore the effects on corticomotor excitability by single low-frequency and high-frequency repetitive transcranial magnetic stimulation. Participants will receive different stimulation approaches in sequences: high-frequency rTMS, low-frequency rTMS, and sham rTMS. They will be randomly assigned to three groups with different stimulation sequences. After each single stimulation, corticomotor excitability, balance, and motor symptoms will be measured. In this study, eighteen PD patients with Hoehn and Yahr stage 1 to 3 will be recruited.
Supporting Information: Study Protocol, CSR, Analytic Code
Time Frame: 5 years